CLINICAL TRIAL: NCT07262177
Title: Mindful Embodied Movement: A 12-Week Modern Dance-Mindfulness Intervention and Mixed-Methods Randomized Controlled Trial in Recreational Adult Dancers
Brief Title: Dance-Mindfulness Intervention for Well-Being in Recreational Adults
Acronym: DanceMind
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Aglaia Zafeiroudi, Academic Staff, Department of Physical Education and Sport Science, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IEC, DPESS, UTH 4-2/2.4.2025; IEC 4-2/2.4.2025 (Other: Department of Physical Education & Sport Science, University of Thessaly, Greece)
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Health Promotion
Keywords: somatic education; embodied phenomenology; community-based dance education; dance movement therapy; psychological wellbeing; mindfulness; creative movement; interoception; autonomic regulation; embodied awareness; emotional regulation; vagal regulation; stress reduction; motor learning
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance-Mindfulness Intervention (Experimental): Participants assigned to the Dance-Mindfulness intervention arm receive 12 weekly sessions (90-100 minutes each) over 12 weeks. Each session integrates: (1) polyvagal-informed breath-movement synchronization, (2) ISTD Modern Theatre Dance technique and dance movements (Grades 2-4), (3) nervous system regulation through somatic practices, and (4) phenomenological reflection via weekly journaling. Sessions follow a standardized 8-component structure with 15-18 participants per session delivered by trained facilitators. Classroom-based, in-person delivery at participating dance schools.
  Interventions: Behavioral: Dance-Mindfulness Intervention
- Control (No Intervention): Participants assigned to the waitlist control arm continue their usual dance activities for 12 weeks, excluding mind-body practices (Pilates, yoga, tai-chi etc). After the 12-week assessment period, all control participants are offered access to the Dance-Mindfulness intervention.

INTERVENTIONS:
Behavioral: Dance-Mindfulness Intervention — A 12-week integrated dance-mindfulness program combining ISTD Modern Theatre Dance technique with polyvagal-informed breathing, somatic practices, and phenomenological reflection. Sessions are 90-100 minutes weekly, delivered in groups of 15-18 participants by trained facilitator(s). The intervention integrates breath-movement synchronization (9-10 min), technical dance work (14-15 min), conditioning (9-10 min), rhythm & improvisation (8-9 min), choreographed sequences (15-17 min), cool-down integration (8-9 min), and phenomenological journaling (10-20 min). Three-phase progression: Phase 1 (Weeks 1-4) establishes safety and foundational skills; Phase 2 (Weeks 5-8) expands embodied exploration; Phase 3 (Weeks 9-12) focuses on expressive integration and self-regulation consolidation.
  Other Names: Mindful Embodied Movement; Modern Dance-Mindfulness Program; ISTD Dance-Mindfulness Integration
  Arms: Dance-Mindfulness Intervention

SUMMARY:
This 12-week study protocol outlines a randomized controlled trial designed to evaluate the effectiveness of a Dance-Mindfulness intervention integrating Modern Theatre Dance with mindfulness-based embodied practices to enhance psychological wellbeing, nervous system regulation, and embodied awareness in adults. The intervention combines: (1) polyvagal-informed breath-movement synchronization (nasal breathing, grounding); (2) ISTD (Imperial Society of Teachers of Dancing) Modern Theatre Dance technique progression and dance movements (Grades 2-4); (3) nervous system regulation through somatic practices; and (4) phenomenological reflection via weekly journaling and post-session integration.

Study Design: Parallel-assignment randomized controlled trial (approx. N=320; n=160 intervention, n=160 waitlist control). Randomization uses computer-generated block randomization (block sizes 4-6).

Outcomes: Perceived stress, mindfulness psychological wellbeing (happiness, life satisfaction), emotional regulation, social connection, movement confidence.

Qualitative Component: Phenomenological interviews and weekly reflective journals from subsample (approx. n=20) analyzed via Interpretative Phenomenological Analysis and Reflexive Thematic Analysis.

Intervention Delivery: 90-100 minute weekly sessions delivered over 12 weeks by qualified facilitator(s) trained in Modern Theatre Dance, mindfulness (≥3 years personal practice, MBSR, yoga or equivalent), trauma-informed care, and group facilitation. Sessions include 8 structured components: breath-grounding (9-10 min), technical dance work (14-15 min), conditioning (9-10 min), break-settling (4-5 min), rhythm improvisation (8-9 min), choreographed sequences (15-17 min), cool-down-integration (8-9 min), and phenomenological journaling (10-20 min).

Safety & Fidelity: Structured facilitator guidelines, session checklists, weekly supervision, adverse event protocols, and external fidelity monitoring ensure protocol integrity. Classroom size: 15-18 participants per session.

Data Collection: Baseline (Week 0), mid-intervention (Week 6 only for qualitative), post-intervention (Week 12), and optional 1-3 month follow-up. Intent to treat analysis and mixed-effects modeling for between-group comparisons. Population: Adults (age 18+) seeking wellbeing enhancement through recreation or stress reduction. Eligible participants without acute mental health crisis. Primary Purpose: Health promotion and mental health improvement through nervous system regulation, embodied awareness, and psychosocial wellbeing enhancement.

DETAILED DESCRIPTION:
This study evaluates a study protocol for a 12-week Dance-Mindfulness intervention designed for recreational adult dancers in community dance schools. The intervention integrates modern dance training with mindfulness, somatic awareness, and polyvagal-informed regulation strategies, applied within an ISTD-based modern theatre dance curriculum. Existing evidence in somatic psychology and embodied movement practices suggests that combining dance with structured mindfulness may enhance emotional regulation, interoceptive awareness, stress reduction, and overall psychological well-being. However, most dance-based interventions occur outside regular dance classes and often target clinical or professional populations. This trial addresses an important gap by implementing a standardized mindfulness-enhanced protocol within routine recreational dance instruction.

Mindfulness practices, including breath regulation and non-judgmental attention to bodily sensations, are associated with improvements in anxiety, mood, and life satisfaction. Dance offers a unique context for embodied learning, combining rhythm, movement sequencing, creative expression, and social interaction. The Dance-Mindfulness protocol integrates these elements to support autonomic regulation, grounding, and embodied awareness during dance practice. Polyvagal principles related to safety, vagal tone, and co-regulation inform specific breathing patterns and pacing. The intervention is structured to enhance psychological engagement with dance, promote meaning-making through movement, and support sustained focus, thus linking contemplative practices with artistic training.

Participants allocated to the intervention attend one weekly session (90-100 minutes) over 12 weeks. Sessions follow a structured curriculum with three progressive phases:

Foundations (Weeks 1-4): grounding practices, breath awareness, interoceptive techniques, and gentle preparatory movement.

Embodied Exploration (Weeks 5-8): integration of ISTD syllabus exercises with mindful pacing, sensory modulation, and guided improvisation.

Expressive Integration (Weeks 9-12): creative tasks, choreography, reflective processes, and strategies for self-regulation during movement.

Each session includes a combination of somatic exercises, mindful movement sequences, modern dance technique, creative exploration, and brief reflective journaling. Instruction is invitational, supporting autonomy, choice, and safety. Environmental conditions (e.g., floor safety, sound levels, lighting) follow standardized preparation procedures across all participating studios to ensure consistent implementation.

Participants assigned to the control group continue their usual dance activities for 12 weeks. Activities that incorporate explicit mindfulness or mind-body components (e.g., yoga, Pilates, tai chi) are excluded during the study period. Control participants do not receive any mindfulness training. After completion of post-intervention assessments, they are offered access to the Dance-Mindfulness program.

All eligible participants complete baseline assessments before randomization (T0) and post-intervention assessments at Week 12 (T2). Measures include psychological well-being, mindfulness, happiness, stress, anxiety, depression, and psychological involvement in dance. These standardized instruments are administered on paper by the site coordinator. A subset of participants provides qualitative data through semi-structured interviews and weekly reflective journaling to explore perceived changes in embodiment, emotional awareness, and personal meaning related to dance. Interviews occur after Week 12 using a structured guide.

To ensure consistency across dance schools, facilitators use a standardized Intervention Manual. Fidelity is supported through session checklists, facilitator notes, and occasional independent observations. All facilitators hold appropriate qualifications in dance teaching, mindfulness-based methods, and safe movement instruction.

The intervention is low-risk and consistent with activities typical in recreational dance settings. Potential physical risks include mild fatigue or muscle soreness. Psychological risks are minimal but may include temporary emotional discomfort associated with contemplative practices. Participants may pause or withdraw at any time. Any adverse events are documented and reported according to institutional guidelines.

This trial aims to determine whether integrating mindfulness into recreational dance practice improves psychological well-being, enhances mindfulness and happiness, reduces stress and negative mood states, and increases psychological engagement with dance. The qualitative component seeks to deepen understanding of how participants experience embodied awareness, emotional regulation, and meaning-making throughout the 12-week process. The study will contribute new evidence regarding mindfulness-based movement interventions in non-clinical adult populations and within naturalistic community dance settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Enrolled in dance classes (preferring modern/contemporary) at participating schools for at least 6 months prior to study enrollment
* Able and willing to attend weekly sessions for 12 consecutive weeks (minimum 70% attendance required)
* Able to understand and complete study questionnaires in Greek language
* Able to engage in moderate-intensity movement and dance activities without acute medical contraindications
* Written informed consent provided
* Willing to be randomly assigned to intervention or waitlist control group

Exclusion Criteria:

* Musculoskeletal or neurological conditions limiting safe participation in moderate-intensity movement (e.g., acute injury, severe arthritis, neurological disease affecting coordination/balance)
* Current severe psychological distress or mental health crisis requiring immediate clinical intervention (screened via DASS-21; cutoff: Severe or Extremely Severe on any subscale)
* Pregnancy or planning pregnancy during the 12-week study period
* Current concurrent participation in other psychological interventions, therapy, or mind-body programs (Pilates, yoga, tai-chi, other mindfulness-based interventions)
* Unable to attend ≥70% of weekly sessions due to scheduling constraints or anticipated absences
* Inability to provide informed consent or complete questionnaires in Greek
* Acute medical illness or hospitalization within 2 weeks of study start
* History of substance abuse disorder currently active or untreated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Life Satisfaction (Satisfaction With Life Scale - SWLS) | Baseline (Week 0) and Post-intervention (Week 12)
  The Satisfaction With Life Scale (SWLS) is a 5-item self-report measure assessing global life satisfaction. Items are rated on a 7-point Likert scale (1 = Strongly Disagree, 7 = Strongly Agree). Total score ranges 5-35, with higher scores indicating greater life satisfaction. Scoring: 31-35 = High satisfaction, 26-30 = Moderate satisfaction, 21-25 = Low satisfaction, 15-20 = Dissatisfied, 5-14 = Highly dissatisfied. The scale has demonstrated reliability (α = .79) and validity across diverse populations. Administration time: 2-3 minutes.
Psychological Distress (DASS-21: Depression, Anxiety, Stress Scale) | Baseline (Week 0) and Post-intervention (Week 12)
  The DASS-21 is a 21-item self-report scale measuring depression, anxiety, and stress across three 7-item subscales. Items are rated 0-3 (0 = Never, 3 = Almost Always). Subscale scores range 0-21 each, with higher scores indicating greater symptom severity. Interpretation per subscale: 0-7 = Normal/Minimal, 8-9 = Mild, 10-14 = Moderate, 15-19 = Severe, 20-21 = Extremely Severe. The scale demonstrates good internal consistency (α = .81-.87 across subscales) and has been validated in Greek populations. Subscales measure: Depression (emotional dysphoria, hopelessness), Anxiety (autonomic arousal, fear, worry), and Stress (tension, irritability, difficulty relaxing). Administration time: 5-7 minutes.
Mindfulness (Mindful Attention Awareness Scale - MAAS) | Baseline (Week 0) and Post-intervention (Week 12)
  The Mindful Attention Awareness Scale (MAAS) is a 15-item unidimensional measure of trait mindfulness, assessing the ability to maintain present-moment attention and awareness. Items are rated on a 6-point Likert scale (1 = Almost Always, 6 = Almost Never). Total scores range 15-90, with higher scores indicating greater mindfulness capacity and present-moment awareness. Interpretation: 15-40 = Low mindfulness, 41-65 = Moderate mindfulness, 66-90 = High mindfulness. The scale demonstrates good internal consistency (α = .82) and has been validated cross-culturally. MAAS captures the core mechanism of mindfulness-based interventions attentional awareness in daily life. Administration time: 4-5 minutes.
Subjective Happiness (Subjective Happiness Scale - SHS) | Baseline (Week 0) and Post-intervention (Week 12)
  The Subjective Happiness Scale (SHS) is a brief 4-item self-report measure of overall happiness and positive affect. Items use varied response formats with 7-point scales. Total scores range 4-28, with higher scores reflecting greater happiness. Interpretation: 4-10 = Unhappy, 11-18 = Moderately happy, 19-28 = Very happy. The scale has demonstrated good reliability (α = .86) and validity as a global well-being indicator. Direction: Higher scores on this measure are desirable and indicate better psychological well-being. Administration time: 2-3 minutes.
Leisure Involvement (Leisure Involvement Scale) | Baseline (Week 0) and Post-intervention (Week 12)
  The Leisure Involvement Scale is a 13-item self-report measure assessing the depth of psychological engagement, personal meaning, and commitment to recreational activities. Items examine dimensions including: activity attractiveness/interest, centrality to life, and personal identity/self-identification through the activity. Participants rate each item on a 7-point Likert scale (1 = Strongly Disagree, 7 = Strongly Agree). Total scores range 13-91, with higher scores indicating greater psychological involvement, personal meaning-making, and identification with recreational dance participation. Direction: Higher scores are desirable and reflect greater embodied engagement, movement identity development, and psychological investment in leisure. The scale has demonstrated reliability and validity for assessing leisure involvement in Greek populations (Theodorakis, Panopoulou, & Vlachopoulos, 2007). Administration time: 5-7 minutes.

SECONDARY OUTCOMES:
Movement Identity and Personal Meaning-Making (Qualitative Narrative Analysis) | Weekly journals (Weeks 1-12); Post-intervention interviews (Week 12)
  Qualitative analysis of journal entries and interviews examining personal meaning-making, movement identity development, and psychological integration of embodied practices. Coded dimensions include: (1) Movement Identity, shifts in self-perception as a mover, dancer, embodied being; changes in body image, movement confidence, creative expression; (2) Meaning-Making, personal significance attributed to dance experience, psychological insights, transformative moments; (3) Life Integration, application of embodied awareness and regulation skills beyond dance sessions; sustained practice and internalization; (4) Social Connection, experienced sense of belonging, group attunement, relational aspects of embodied practice. Qualitative meaning-making themes complement quantitative leisure involvement and life satisfaction outcomes, illustrating the depth of psychological and identity-level changes fostered by the integrated Dance-Mindfulness program.

CONTACTS AND LOCATIONS:
Overall Officials: Aglaia Zafeiroudi, SES, Study Chair — University of Thessaly; Charilaos Kouthouris, Study Director — University of Thessaly; Aglaia Zafeiroudi, SES, Principal Investigator — University of Thessaly
Locations (1):
- Department of PE and Sport Science (DPESS), University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No